CLINICAL TRIAL: NCT01811537
Title: Phase II Study of Using a New Device (Neochordameter) in Making Artificial Chordae for Mitral Valve Repair
Brief Title: Safety and Efficacy Study of a New Device for Making Neochordae in Mitral Valve Repair
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Alireza Ghavidel, Associat Professor of Cardiac Surgery, Tehran University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 91-01-149-17122-59685
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Mitral Valve Repair
Keywords: Artificial Chordae; Mitral Valve Repair

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental: premeasured Neochordae (Experimental): Transthoracic echocardiography(TTE) is done for all patients. The new device will be setup using the TTE measurements.The artificial Chordae loops will be made at the operation room before starting the surgery. These loops will be attached to the respective papillary muscle's head and the free edge of respective prolapsed scallop.
  Interventions: Device: Artificial Chordae

INTERVENTIONS:
Device: Artificial Chordae

SUMMARY:
Mitral prolapse is a common cardiac disease whose patients are at higher risk for serious complications. Mitral valve (MV) repair offers several important advantages compared with valve replacement and it achieves excellent midterm and long-term results. Two major problems of using pre-measured expanded polytetrafluoroethylene(ePTFE) neochordae (the loop technique) are deciding the length of the neochordae and tying the knot at the intended length. Therefore, a great need still exists to find new method to simplify and precise the length of neochordae. 20 patients with mitral valve prolapse who undergo mitral valve repair using neochorda will be recruited in this study. Trans thoracic echocardiography (TTE) will be done preoperatively for all patients. Two, three, and four chamber view of each patient will be pre-operatively recorded. The device will be set with extracted measurements. Artificial corda loops are made using CV-4 ePTFE sutures. After artificial chordae replacement, the ring annuloplasty will be done. Follow up: A leakage test after attaching the 1st loop; Post operative trans esophageal echocardiography (TEE) and determining the severity of mitral regurgitation [Wall motion Score Index (WMSI), Mitral Annulus Area (MAA), LVEF, End Systolic Volume (ESV), End Diastolic Volume (EDV), Iso-Volemic Relaxation Time (IVRT), (IVRT/(QE-QE^') ,Chamber Relaxation velocity)/(Myocard relaxation velocity(E/E^' ), HR]; TEE 3 months after discharge; Cross clamp time; Intubation period in ICU.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Mitral valve prolapse who undergo mitral valve repair using neochorda

Exclusion Criteria:

* Nothing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Mortality | Early (within 30 days after surgery), Late (After 12 months)

SECONDARY OUTCOMES:
Mitral Valve prolapse measurement after using neochordae | Intra-operation, 3, 6, and 12 months after surgery

OTHER OUTCOMES:
Cardiopulmonary bypass time | During Surgery